CLINICAL TRIAL: NCT02758821
Title: The Impact of C-reactive Protein Testing on Antibiotic Prescription in Febrile Patients Attending Primary Care in Low-resource Settings
Brief Title: The Impact of C-reactive Protein Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Department of Medical Research, Lower Myanmar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CRP POC
Record Dates: First submitted 2016-03-10; First posted 2016-05-03 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Fever
Keywords: C-reactive protein; antibiotic
MeSH Terms: conditions — Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRP-Control (Other): The health care provider will manage the patient using standard guidelines. No CRP will be measured onsite
  Interventions: Other: No CRP will be measured onsite
- CRP-A (Other): CRP will be measured by a study nurse onsite and the result will be communicated to the health care provider.
  Interventions: Other: CRP cut-off of 20mg/L.
- CRP-B (Other): CRP will be measured by a study nurse onsite and the result will be communicated to the health care provider.
  Interventions: Other: CRP cut-off of 40mg/L.

INTERVENTIONS:
Other: No CRP will be measured onsite — No CRP will be measured onsite
  Arms: CRP-Control
Other: CRP cut-off of 20mg/L. — Health care worker will be given an advice to prescribe antibiotic to patient who has CRP lever < 20mg/L.
  Arms: CRP-A
Other: CRP cut-off of 40mg/L. — Health care worker will be given an advice to prescribe antibiotic to patient who has CRP lever < 40mg/L.
  Arms: CRP-B

SUMMARY:
PRIMARY OBJECTIVE To assess the impact of C-reactive protein (CRP) Point-of-care (POC) testing on health care worker prescribing behaviour in patients presenting to primary healthcare centres with an acute fever or recent history of fever.

SECONDARY OBJECTIVES To assess the impact of CRP testing on clinical outcomes within the 14 days of follow-up.

To assess the correlation between CRP results and clinical outcomes on the day 5 of the enrolment.

To estimate the impact of CRP testing on antibiotic consumption after first consultation.

To explore the attitudes of health centre staff towards the POC CRP test. To identify the prevalence of key pathogens in febrile patients in these settings.

To validate the ability of CRP to discriminate between viral and bacterial pathogens in a subset of patients with a microbiologically confirmed diagnosis.

DETAILED DESCRIPTION:
This is a multi-centre, individually randomized-controlled, three-armed pragmatic trial comparing CRP guided antibiotic prescription in febrile patients to the current standard prescribing systems. The study will be implemented in low and middle-income countries in tropical settings, including Myanmar and Thailand in the first instance.

As participation in the study itself may raise awareness amongst the health centre staff and local community, current antibiotic prescribing rates will be assessed in an observational run-in period before the intervention. Health workers will be asked to complete case record forms (CRF) for patients presenting to their health centre with current or recent fever. This aims to capture current antibiotic prescribing habits before the study is launched.

During the intervention phase, patients fulfilling the inclusion criteria and who consent to participate in the study will be randomised to one of the three arms, as follows:

1. Control group: The health care provider will manage the patient using standard guidelines. No CRP will be measured onsite
2. Group A: CRP will be measured by a study nurse and the result will be communicated to the health care provider as "High-CRP" or "Low-CRP" using a low CRP cut-off of 20mg/L.
3. Group B: CRP will be measured by a study nurse and the result will be communicated to the health care provider as "High-CRP" or "Low-CRP" using the higher CRP cut-off, of 40mg/L.

For the two intervention arms, the following guidance will be given to the health care provider: if the CRP test is reported as 'high', antibiotic treatment is recommended, following local guidelines, and if it is reported as 'low' antibiotics are not recommended. In either case the information provided by the CRP test should be interpreted alongside their clinical judgement.

A second CRP will be sampled at day 5 of the follow-up (+/- 1 day) for all the patients, using capillary blood from a finger prick.

The investigators will use the NycoCard Reader II (Axis Shield, Norway or equivalent) to measure CRP levels.

A venous blood sample and a nasopharyngeal swab will be taken in the control group at enrolment and sent to a central laboratory in order to detect the presence of the following key pathogens by real-time polymerase chain reaction (PCR):

* Flavivirus
* Alphavirus
* Influenza A & B
* Rickettsia including typhus group and spotted fever group
* Leptospirosis
* PCR 16s for the detection of any bacteria.
* Malaria

CRP will also be retrospectively measured in these blood samples to validate its ability to distinguish between viral and bacterial infections.

A urine sample will be collected to detect the presence of antimicrobials at day 0 and day 5. This procedure will ascertain pre-study antibiotic intake, as well as the patient's compliance to the health care worker's prescription or advice that antibiotics are not required, during their participation in the study. The urine samples will be collected at the sites, divided into aliquots and frozen to -80°c to be stored on site. Monthly shipments will be made to the laboratory at Mahidol Oxford Tropical Research Medicine Unit in Thailand for analysis.

The investigators aim to follow-up every patient face to face on day 5 (+/-1 day), and either by phone or face-to-face interviews 14 days (+/-2 days) after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥1 year presenting to selected primary healthcare centres
* Tympanic temperature >37.5°c or history of fever ≤ 14 days.

Exclusion Criteria:

* Patients that in view of the study nurse are in need of emergency referral to a higher-level facility, as indicated by either 1) impaired consciousness or 2) inability to take oral medication.
* In sites that routinely test for malaria, patients with a positive malaria rapid diagnostic test or microscopy will be excluded
* The main complaint is a trauma and/or injury
* Suspicion of tuberculosis (any medical history and/or physical examination suggesting tuberculosis)
* Suspicion of Urinary Tract Infections (any medical history and/or physical examination suggesting urinary tract infections)
* Suspicion of local skin/dental abscess (any medical history and/or physical examination suggesting a local skin/dental abscess
* Any presenting symptom present for more than 14 days
* Bleeding, including otorrhagia, haematemesis, haemoptysis, haemorrhagic petechiae, haematuria, bloody diarrhoea.
* Not able to comply with the follow-up at Day 5 (+ / - 1 day).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2410 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The proportion of recruited patients prescribed an antibiotic | 6 Days
  The proportion of recruited patients prescribed an antibiotic at the health centre on or between their enrolment and the first follow-up visit (on day 5 +/- 1 day).

SECONDARY OUTCOMES:
Duration of symptoms | 14 Days
  Symptoms as defined by fever, any other symptom
Severity of symptoms | 14 Days
  Severity will be assessed by the nurse using a rating scale graded from 1 to 4 (#Grading 1=mild, 2=moderate, 3=severe, 4=potentially life-threatening), according to the patients' description of their symptoms, and the findings of the physical examination.
Frequency of severe clinical outcomes | 14 Days
  as defined by admission to hospital or death within the 14 days of follow up
Proportion of patients that needed their clinical management changed within the 14 days of follow-up. | 14 Days
Frequency of unplanned re-consultation | 14 Days
Clinical outcome on Day 5 compare to CRP level | 5 Days
Proportion of patients with an immediate versus subsequent prescription within 2 weeks. | 14 Days
Proportion of urine samples that tested positive for presence of antibiotics | 14 Days
Interview of health centre staff for attitudes and satisfaction | 6 months
  Attitudes and satisfaction of health centre staff towards the CRP POC test
The proportion of a population who have key pathogens | 6 months
  Key pathogens are Flavivirus, Alphavirus, Influenza A & B, Rickettsia including typhus group and spotted fever group, Leptospirosis, PCR 16s for the detection of any bacteria and malaria
Percentage of subjects who are correctly identified as having bacterial infections by using CRP testing | 6 months
  Sensitivity is defined as the proportion of patients with high CRP, out of all PCR confirmed bacterial infections.
Percentage of subjects who are correctly identified as having viral infections by using CRP testing | 6 months
  Specificity is defined as the proportion of patients with low CRP, out of all PCR confirmed viral infections.
The likelihood ratio (LR) of correctly identifying a bacterial infection by using CRP-testing. | 6 months
  The positive likelihood ratio is the fraction of sensitivity over (1 - Specificity) , and the negative likelihood ratio is the fraction of (1 - Sensitivity) over Specificity.
The receiver operating characteristic (ROC) for evaluating the accuracy of CRP-testing in identifying bacterial infections. | 6 months
  We will use the ROC, or ROC curve, as a graphical plot, in order to illustrate the performance of the CRP-testing to classify bacterial and non-bacterial infections as its discrimination threshold is varied.

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Lubell, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chiangrai Clinical research Unit, Chiangrai, Chiangrai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Althaus T, Thaipadungpanit J, Greer RC, Swe MMM, Dittrich S, Peerawaranun P, Smit PW, Wangrangsimakul T, Blacksell S, Winchell JM, Diaz MH, Day NPJ, Smithuis F, Turner P, Lubell Y. Causes of fever in primary care in Southeast Asia and the performance of C-reactive protein in discriminating bacterial from viral pathogens. Int J Infect Dis. 2020 Jul;96:334-342. doi: 10.1016/j.ijid.2020.05.016. Epub 2020 May 11. PMID 32437937
- [Derived] Haenssgen MJ, Charoenboon N, Do NTT, Althaus T, Khine Zaw Y, Wertheim HFL, Lubell Y. How context can impact clinical trials: a multi-country qualitative case study comparison of diagnostic biomarker test interventions. Trials. 2019 Feb 8;20(1):111. doi: 10.1186/s13063-019-3215-9. PMID 30736818
- [Derived] Althaus T, Greer RC, Swe MMM, Cohen J, Tun NN, Heaton J, Nedsuwan S, Intralawan D, Sumpradit N, Dittrich S, Doran Z, Waithira N, Thu HM, Win H, Thaipadungpanit J, Srilohasin P, Mukaka M, Smit PW, Charoenboon EN, Haenssgen MJ, Wangrangsimakul T, Blacksell S, Limmathurotsakul D, Day N, Smithuis F, Lubell Y. Effect of point-of-care C-reactive protein testing on antibiotic prescription in febrile patients attending primary care in Thailand and Myanmar: an open-label, randomised, controlled trial. Lancet Glob Health. 2019 Jan;7(1):e119-e131. doi: 10.1016/S2214-109X(18)30444-3. PMID 30554748